CLINICAL TRIAL: NCT06871254
Title: Spinal Cord Injury Neurorecovery Collaboration (SCINC) Master Protocol
Brief Title: Spinal Cord Injury Neurorecovery Collaboration
Acronym: SCINC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Melbourne (Other)
Collaborators: Institute of Breathing and Sleep (Unknown); Austin Health (Other Government); Neuroscience Research Australia (Other); The University of New South Wales (Other); University of Sydney (Other); University of Florida (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCINC_MASTER
Record Dates: First submitted 2025-02-27; First posted 2025-03-11 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-02

CONDITIONS: Spinal Cord Injuries
MeSH Terms: conditions — Spinal Cord Injuries | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Adaptive design Master Protocol investigating multiple interventions within multiple study-specific Appendices.
Masking Description: SCINC Master protocol:
  - Where multiple simultaneous appendices/interventions are evaluated the intent is to keep the independent assessor blinded to the intervention allocation.
  RRULI: Appendix 1:
  - The outcome assessor will be independent of the providers of therapy.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- RRULI: Appendix 1 (Experimental): In this first arm of SCINC, adults with chronic tetraplegia will be assigned to the RRULI: Appendix 1 intervention.
  Interventions: Other: Therapeutic Intermittent Hypoxia (TIH) + Exercise Training (ET)

INTERVENTIONS:
Other: Therapeutic Intermittent Hypoxia (TIH) + Exercise Training (ET) — TIH in combination with upper limb and respiratory ET. The intervention is predominantly home-based and will be delivered three times per week for six weeks.
  Other Names: Therapeutic acute intermittent hypoxia (tAIH); Acute intermittent hypoxia (AIH)

SUMMARY:
SCINC is an adaptive design Master protocol that seeks to determine if there is "sufficient promise" of beneficial effect of treatment combinations to enhance motor recovery in pre-specified strata of people with a spinal cord injury.

DETAILED DESCRIPTION:
SCINC utilises an adaptive design with interim analyses to assess whether a given intervention is futile or shows a "signal of benefit" within an appendix-specific study. The SCINC Master Protocol describes trial procedures, data collection, data monitoring, follow-up visits, and safety procedures that will be employed in all study-specific Appendices. The study-specific Appendix is a Bayesian optimised phase IIA trial, operating under the overarching SCINC Master Protocol. The first study-specific appendix is: Restoration of Respiratory and Upper Limb function after cervical spinal cord Injury (RRULI): Therapeutic Intermittent Hypoxia (TIH) + Exercise Training (ET). The RULLI: Appendix 1 (TIH + ET) aims to determine if ET plus TIH in people with chronic tetraplegia is a therapy with sufficient promise to test in a Phase IIb/III trial; considering feasibility, safety and efficacy. As new interventions are put forth, they will be added to the Master Protocol as a new Appendix. This Master Protocol describes trial procedures, data collection, data monitoring, follow-up visits, and safety procedures that will be employed in all study-specific Appendices. Each study-specific Appendix will have a process evaluation protocol.

ELIGIBILITY:
SCINC Inclusion Criteria:

- Person with SCI

SCINC Exclusion Criteria:

- Proven contraindication to intervention

RRULI: Appendix 1 (TIH + ET) study-specific inclusion criteria:

* Adults > 18 years of age
* Able to independently ventilate
* Chronic SCI (>1 years post-injury or impairment onset)
* Tetraplegia (C2-T1 level of injury)
* Evidence of motor incomplete paralysis in the upper limb below the neurological level of injury
* Have a documented management plan for their AD if it occurs.

RRULI: Appendix 1 (TIH + ET) study-specific exclusion criteria:

* Pregnancy
* Medical instability, including current or recent (within the previous 6 weeks) infection or inflammation
* Current or recent (within the previous 6 weeks) pressure ulcers or cutaneous lesions
* Poorly controlled diabetes
* An episode of AD in the previous 6 months that required medical intervention to resolve
* Significant other neurological, psychiatric, pulmonary, cardiovascular, orthopaedic, or oncological conditions.
* Currently taking part in another clinical trial
* Upper limb contracture

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
At an individual participant level, the Phase IIA study has a single, binary, composite primary outcome to determine if there is a 'signal of benefit', measuring effectiveness, no deterioration, safety and acceptability. | Baseline and 6-weeks.
  The single binary outcome includes the following components:
  A) Effectiveness - Increase above baseline that is equal or more than the predefined outcome-specific stated thresholds, on at least ONE of the: Action Reach Arm Test (ARAT), Handheld dynamometer (GRIP) Maximal inspiratory pressure (MIP) B) No deterioration - No deterioration below baseline. C) Safety - Incidence of Autonomic Dysreflexia (AD) episodes occurring during the intervention period for each individual participant.
  D) Acceptability - Rate of participant adherence to intervention sessions. Please refer to the following primary outcomes for details of each of these components.
A) Effectiveness: Increase above baseline that is equal or more than the predefined outcome-specific stated thresholds, on at least ONE of the: Action Reach Arm Test (ARAT), Handheld dynamometer (GRIP) Maximal inspiratory pressure (MIP) | Baseline and 6 week follow-up
  ARAT: Assesses grasp, grip, pinch and gross movement. A minimal clinically important difference of 5.7 points is accepted in SCI.
  GRIP: Grip strength will be measured according to a standardised procedure. A threshold of 5.0 kg will be used.
  MIP: Respiratory muscle strength will be measured according to standard procedures. A threshold of 10cmH20 will be used.
B) No deterioration | Baseline and 6 week follow-up
  No deterioration (decline below baseline) that is equal or more than the predefined outcome-specific stated threshold, on ANY of the ARAT, GRIP and MIP.
C) Safety - Incidence of Autonomic Dysreflexia (AD) episodes occurring during the intervention period for each individual participant. | Up to 6 weeks.
  Fewer than two AD events that fail to resolve with participants usual, community interventions.
D) Acceptability - Rate of participant adherence to the intervention, as assessed by monitoring attendance to treatment sessions.. | Up to 6 weeks.
  Adherence with at least 70% of treatment sessions.

SECONDARY OUTCOMES:
9-hole Peg test | Baseline and 6-weeks.
  A test of upper limb dexterity and function. This test will be undertaken using the dominant hand.
Pinch grip dynamometer | Baseline and 6-weeks.
  Pinch strength
Penn Spasm Frequency Scale | Baseline and 6-weeks.
  Self-report measure of upper limb spasticity composed of 2-parts:
  1. Spasm frequency: scale 0 (no spasm) - 4 (spasms occurring more than 10 times per hour).
  2. Spasm severity: scale 1 (mild) - 3 (severe). A higher score indicates a worse outcome for both components of the scale.
Capabilities of upper extremity questionnaire | Baseline and 6 weeks
  Questionnaire assessing upper limb function. Scored on a 7-point scale representing self-perceived difficulty:
  1= "totally limited, can't do at all" 7= "not at all limited" Minimum score = 32 Maximum score = 224 (higher score = greater function)
Sleep quality and Obstructive Sleep Apnoea (OSA) will be assessed using polysomnography (a sleep study) | 1 day
  In the week prior to the intervention period, a home-based overnight polysomnography test will occur in the participants home to assess for OSA.
Perceived work of breathing | Baseline and 6-weeks.
  Modified Borg dyspnoea scale. A scale from 0 (no difficulty breathing) - 10 (very, very severe) - where a higher score is a worse outcome.
Respiratory function will assessed using spirometry. | Baseline and 6-weeks.
  Respiratory function measurement - physiological. Spirometry is a test of lung function and can measure how much air a person can force out of their lungs in 1 second (FEV1), and in total (forced vital capacity, FVC).
Maximal expiratory pressure (MEP) and sniff nasal inspiratory pressure (SNIP) | Baseline and 6-weeks
  Respiratory muscle strength
Peak cough flow (L/min) | Baseline and 6-weeks
  Cough effectiveness
Minute Ventilation (Litres) | Baseline and 6-weeks.
  Ventilation response measurement - physiological.
End of tidal breathing oxygen and carbon dioxide saturation. | Baseline and 6-weeks.
  Ventilation response measurement - physiological.
Respiratory Rate measured in breaths per minute. | Baseline and 6-weeks.
  Ventilation response measurement - physiological.
Tidal volume, measured in litres. | Baseline and 6-weeks.
  Ventilation response measurement - physiological measure.
Ventilation response - assessing mouth pressure (measured in cmH20) | Baseline and 6-weeks.
  Ventilation response measure - physiological.
Inspiratory time, measured in seconds (s). | Baseline and 6-weeks.
  Ventilation response measurement - physiological.
Inspiratory and expiratory flow, measured in Litres per second (L/s). | Baseline and 6-weeks.
  Ventilation response measurement - physiological.

CONTACTS AND LOCATIONS:
Overall Officials: David Berlowitz, PhD, Principal Investigator — University of Melbourne
Locations (1):
- Austin Health, Heidelberg, Victoria, Australia

IPD SHARING:
Plan to Share IPD: Yes
De-identified participant level data will be made available for research purposes upon approval of written requests at completion of the trial.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Unending - beginning nine months following publication with no end date.
Access Criteria: Proposals to access IPD must be directed to the study-specific principal investigator.